CLINICAL TRIAL: NCT04304950
Title: Chronotherapy in Inflammatory Bowel Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Garth Swanson, MD, Associate Professor of Medicine Director, Rush Center of Crohn's & Colitis Director, Clinical Chronobiology Center, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16040505
Record Dates: First submitted 2019-08-06; First posted 2020-03-12 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups: Evening Time or Morning Time. Participants are used as their own control. The evening time group will take their medication in the evening and the morning time group will take the medication in the morning.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning (Experimental): Participants with Ulcerative Colitis or Crohn's Disease taking 6-Mercatopurine or Azathioprine orally once a day in the evening were assigned to the morning group. Instead of taking their medication at their usual PM time, they were instructed to take their medications in the morning for the duration of the study-10 weeks. The dosage amount is per clinical care and not defined by the study protocol.
  Interventions: Drug: Morning Group
- Evening (Experimental): Participants with Ulcerative Colitis or Crohn's Disease taking 6-Mercatopurine or Azathioprine orally once a day in the morning were assigned to the evening group. Instead of taking their medication at their usual AM time, they were instructed to take their medications in the evening for the duration of the study-10 weeks. The dosage amount is per clinical care and not defined by the study protocol.
  Interventions: Drug: Evening Group

INTERVENTIONS:
Drug: Evening Group — Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 pm and 11:00 pm.
  Arms: Evening
Drug: Morning Group — Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 am and 11:00 am.
  Arms: Morning

SUMMARY:
This study aims to determine if there is any difference in the efficacy of Inflammatory Bowel Disease (IBD) medication and disease outcomes when taken in the morning or in the evening. The IBD medications being observed are azathioprine and 6-mercaptopurine. The study team believes that there may be a benefit to taking the medication at a certain time of day. To test this theory the study asks participants who are already taking either azathioprine or 6-mercaptopurine for IBD to take the medication consistently at either the morning or in the evening based on when they currently take their medication. Participation is up to 10 weeks +/- 3 days. There will be 2 study visits where the participant will be asked to fill in questionnaires related to their IBD symptoms, their sleep habits, sleep quality, and general health information followed by a blood draw.

DETAILED DESCRIPTION:
The objective of this study is to determine whether the timing of drug administration to treat inflammatory bowel disease (IBD) has an effect on patient outcomes. Primary objective: Determine whether there is a difference in outcomes seen when patients are assigned to take their prescribed immunomodulator (IM) - either Azathioprine or 6-Mercaptopurine - at either a morning delivery time or evening delivery time.

The Investigator hypothesize that administration time of immunomodulators (IMs) during the day can affect the clinical outcomes in IBD patients.

Specific Aims Include:

* Determine whether morning vs. evening dosing of patients' prescribed IMs (either Azathioprine or 6-Mercaptopurine) could affect the subclinical markers of inflammation related to disease.
* Determine whether morning vs. evening dosing of patients' prescribed IMs (either Azathioprine or 6-Mercaptopurine) could affect endoscopic outcomes.
* Determine whether morning vs. evening dosing of IMs affect their biochemical side effects, as is routinely monitored as part of the patients' clinical care.
* Determine if outcomes correlate with patients' chronotype, as determined by standard questionnaires (the Munich Chronotype Questionnaire).

Description of Procedures: After signing the informed consent form, subjects will be asked to answer the Inflammatory Bowel Disease Questionnaire (IBDQ), the Munich Chronotype Questionnaire (MCTQ), the Harvey Bradshaw questionnaire, and a demographics survey. All six of these questionnaires are included with this IRB. Next, patients will be assigned a time (morning or evening) to self administer their prescribed medication for 10 weeks. Patients who currently take their medication in the morning will be asked to switch to an evening delivery and patients who currently take their medication at night will be asked to switch to a morning delivery. The group assigned to morning delivery time will be told to take their medication between 6am and 11am. The group assigned to evening delivery time will be told to take their medication between 6pm and 11pm. Lastly, patients will be asked to give a blood sample to test for complete blood count (CBC), comprehensive metabolic panel (CMP), C-reactive protein (CRP), methylmercaptopurine (6-MMP), and thioguanine nucleotides (6-TG). Plasma and serum isolated from the blood sample will be temporarily stored to measure inflammatory cytokines after every 20 subjects complete the study.

Within a 6-10 week window, as part of their clinical care, subjects will come in to assess their clinical status while undergoing biochemical monitoring every 2-4 weeks. Data from their endoscopic examination, if done, will also be collected.

After 10 weeks, the subjects will be asked to complete the IBDQ and Harvey Bradshaw questionnaire. In addition, a blood sample will be obtained to measure the same metabolite levels and other biochemical indications of disease as stated above. Again, plasma and serum will be isolated from the blood sample and stored.

ELIGIBILITY:
Inclusion Criteria:

* Above the ages of 18
* Diagnosis of Crohn's Disease or Ulcerative Colitis
* Currently taking azathioprine or 6-mercaptopurine
* Willing to sign study consent form

Exclusion Criteria:

* Vulnerable population (pregnant, prisoner, non-English speaking or cognitively impaired)
* Breastfeeding subject
* Have a history of complications related to immunomodulatory therapy
* Participating in other research studies involving research interventions
* Treated with dual corticosteroid and immunomodulatory therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2023-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garth Swanson, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ardizzone S, Bianchi Porro G. Biologic therapy for inflammatory bowel disease. Drugs. 2005;65(16):2253-86. doi: 10.2165/00003495-200565160-00002. PMID 16266194
- [Background] Belaiche J, Desager JP, Horsmans Y, Louis E. Therapeutic drug monitoring of azathioprine and 6-mercaptopurine metabolites in Crohn disease. Scand J Gastroenterol. 2001 Jan;36(1):71-6. doi: 10.1080/00365520150218084. PMID 11218242
- [Background] Bradford K, Shih DQ. Optimizing 6-mercaptopurine and azathioprine therapy in the management of inflammatory bowel disease. World J Gastroenterol. 2011 Oct 7;17(37):4166-73. doi: 10.3748/wjg.v17.i37.4166. PMID 22072847
- [Background] Grevenitis P, Thomas A, Lodhia N. Medical Therapy for Inflammatory Bowel Disease. Surg Clin North Am. 2015 Dec;95(6):1159-82, vi. doi: 10.1016/j.suc.2015.08.004. Epub 2015 Oct 23. PMID 26596920
- [Background] Gomez-Gomez GJ, Masedo A, Yela C, Martinez-Montiel Mdel P, Casis B. Current stage in inflammatory bowel disease: What is next? World J Gastroenterol. 2015 Oct 28;21(40):11282-303. doi: 10.3748/wjg.v21.i40.11282. PMID 26525013
- [Background] Haus E, Sackett-Lundeen L, Smolensky MH. Rheumatoid arthritis: circadian rhythms in disease activity, signs and symptoms, and rationale for chronotherapy with corticosteroids and other medications. Bull NYU Hosp Jt Dis. 2012;70 Suppl 1:3-10. PMID 23259651
- [Background] Perri D, Cole DE, Friedman O, Piliotis E, Mintz S, Adhikari NK. Azathioprine and diffuse alveolar haemorrhage: the pharmacogenetics of thiopurine methyltransferase. Eur Respir J. 2007 Nov;30(5):1014-7. doi: 10.1183/09031936.00026107. PMID 17978158
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523
- [Derived] Swanson GR, Biglin M, Raff H, Chouhan V, Jochum S, Shaikh M, Francey L, Bishehsari F, Hogenesch J, Keshavarzian A. Impact of Chronotherapy on 6-Mercaptopurine Metabolites in Inflammatory Bowel Disease: A Pilot Crossover Trial. Clin Transl Gastroenterol. 2023 Feb 1;14(2):e00549. doi: 10.14309/ctg.0000000000000549. PMID 36730289
- See also: Immunomodulators. (2009, January 16). Retrieved from Crohn's & Colitis Foundation of America — https://www.crohnscolitisfoundation.org/what-is-ibd/medication/immunomodulators
- See also: Inflammatory bowel disease. (2014, September 4). Retrieved February 25, 2016, from Centers for Disease Control and Prevention Website — http://www.cdc.gov/ibd/index.htm
- See also: MacDermott, R. P. (2016). 6-mercaptopurine (6-MP) metabolite monitoring and TPMT testingin the treatment of inflammatory bowel disease with 6-MP or azathioprine. RetrievedMarch 6, 2016, from UpToDate website — http://www.uptodate.com/contents/6-mercaptopurine-6-mp-metabolite-monitoring-and-tpmt-testing-in-the-treatment-of-inflammatory-bowel-disease-with-6-mp-or-azathioprine

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to groups based only on morning vs. evening medication administration status, not on their IBD condition or medication. This study focuses on the timing of medication. It was pre-specified in the protocol to report data based on timing. No plans were made to further stratify the data into more groups. After completing the first research visit, all subjects were asked to take their medication at the opposite time of day from their baseline for 10 weeks.
Groups:
- Evening Group Medication Administration: Participants with Ulcerative Colitis or Crohn's Disease taking Azathioprine or 6- Mercaptopurine orally once a day in the morning were assigned to the evening group. Dosage amount is per clinical care and not defined by the study protocol.
  Evening Group: Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 pm and 11:00 pm for the duration of the study (10 weeks).
- Morning Group Administration: Participants with Ulcerative Colitis or Crohn's Disease taking Azathioprine or 6- Mercaptopurine orally once a day in the evening were assigned to the morning intervention group. Dosage amount is per clinical care and not defined by the study protocol.
  Morning Group: Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 am and 11:00 am for the duration of the study (10 weeks)
Period: Overall Study
Arm/Group | Evening Group Medication Administration | Morning Group Administration
Started | 19 | 9
Completed | 18 | 8
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Evening Group Medication Administration: Participants with Ulcerative Colitis taking Azathioprine or 6-Mercaptopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Participants with Crohn's Disease taking Azathioprine or 6-Mercaptopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Evening Group: Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 pm and 11:00 pm.
- Morning Group Medication Administration: Participants with Ulcerative Colitis taking 6-Mercatopurine or 6-Mercaptopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Participants with Crohn's Disease taking Azathioprine or 6-Mercaptopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Morning Group: Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 am and 11:00 am.
- Total: Total of all reporting groups
Arm/Group | Evening Group Medication Administration | Morning Group Medication Administration | Total
Number analyzed (Participants) | 18 | 8 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 9 | 1 | 10
Age, Continuous [Median (Full Range); unit: years] | 64 [24 to 85] | 32.5 [3 to 79] | 57 [3 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 14
  Male | 6 | 6 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 16 | 5 | 21
  African American | 2 | 2 | 4
  Asian | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Thioguanine Levels in Blood (Morning Versus Evening Dosing)
Description: This is to examine if the intervention results in a greater level of thioguanine in the participants. If so, the participants are expected to have less symptom severity. Comparing baseline taken at visit one to visit two levels 10 weeks after intervention start.
Time Frame: 10 weeks post baseline visit.
Population: During the analysis, the PI and study team grouped participants by their AM and PM medication administration, regardless of what condition or medication they were on. UC and CD are types of IBD, so the analysis focuses on timing of medication in IBD. Unable to find and recruit UC patients on 6-MP.
Measure: Mean (Standard Deviation); unit: pmol/8 x 10^8 RBC
Groups:
- Morning Group Medication Administration: Participants with Ulcerative Colitis taking Azathioprine or 6-Mercaptopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Participants with Crohn's Disease taking Azathioprine or 6-Mercaptopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Morning Group: Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 am and 11:00 am.
Arm/Group | Evening Group Medication Administration | Morning Group Medication Administration
Number analyzed (Participants) | 18 | 8
pmol/8 x 10^8 RBC | 175.04 (106.89) | 225.65 (155.05)

2. Primary Outcome: Harvey Bradshaw Activity Index
Description: Harvey Bradshaw Activity Index has 5 questions. The final score is totaled and will fall into the following categories, which are used to define the severity of the disease: >16 severe diseases, 8-16 moderate disease, 5-7 mild disease, <5 remission. Scores range from 0 ( lowest possible score) to 17.
Time Frame: 10 weeks post baseline visit.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Morning Group Medication Administration: Participants with Ulcerative Colitis taking Azathioprine or 6-Mercaptopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Participants with Ulcerative Colitis taking Azathioprine or 6-Mercaptopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Participants with Crohn's Disease taking Azathioprine or 6-Mercaptopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Morning Group: Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 am and 11:00 am.
Arm/Group | Evening Group Medication Administration | Morning Group Medication Administration
Number analyzed (Participants) | 18 | 8
units on a scale | 2.15 (1.71) | 3.09 (2.71)

3. Primary Outcome: Short Inflammatory Bowel Disease Questionnaire
Description: Quality of Life Measure Score:1-7 (The higher the number the greater the quality of life)
Time Frame: 10 weeks post baseline visit.
Population: During the analysis participants were grouped by AM and PM administration. UC and CD are types of IBD. The study team was unable to recruit Ulcerative Colitis individuals on 6-MP as was originally intended.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Evening Group Medication Administration | Morning Group Medication Administration
Number analyzed (Participants) | 18 | 8
units on a scale | 5.83 (0.56) | 5.91 (0.63)

4. Primary Outcome: 6-Methylmercaptopurine Levels in Blood
Description: This is to examine if the intervention results in a lower level of 6-Methylmercaptopurine in the participants. If so, the participants are expected to have less symptom severity. Comparing baseline taken at visit one to visit two levels 10 weeks after intervention start.
Time Frame: 10 weeks post baseline visit.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/8 x 10 ^8 RBC
Arm/Group | Evening Group Medication Administration | Morning Group Medication Administration
Number analyzed (Participants) | 18 | 8
pmol/8 x 10 ^8 RBC | 2395.27 (2880.26) | 825.15 (1023.34)

5. Secondary Outcome: Munich Chronotype Questionnaire ( MCTQ)
Description: This questionnaire is used to collect primary sleep times, such as bed- and rise-times, including the time a person is fully awake, sleep latency and inertia, in addition to other time points. The MCTQ uses the midpoint of sleep between sleep onset and offset to assess chronotype. Chronotype is your body's natural time to be awake or asleep at certain times. Total scores can range from 16 to 86, with the lowest values representing extreme-late chronotype. For this study corrected midpoint of sleep (MSFc) was calculated. This information is combined to determine the mean time of day at which respondents were more likely to feel most alert. The numbers provided in the outcome measure data table represent time (hour and minute). The hour has been converted to military time and the minutes were converted to decimals.
Time Frame: 10 weeks post baseline visit.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Evening Group Medication Administration: Participants with Ulcerative Colitis taking Azathioprine or 6-Mercatopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Participants with Crohn's Disease taking Azathioprine or 6-Mercatopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Evening Group: Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 pm and 11:00 pm.
- Morning Group Medication Administraion: Participants with Ulcerative Colitis taking Azathioprine or 6-Mercatopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Participants with Crohn's Disease taking Azathioprine or 6-Mercatopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Morning Group: Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 am and 11:00 am.
Arm/Group | Evening Group Medication Administration | Morning Group Medication Administraion
Number analyzed (Participants) | 18 | 8
hours | 3.70 (1.09) | 2.57 (1.21)

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Description: Participants were monitored throughout the study and an adverse events log was kept. However, there are no major risks or discomforts associated with this study. The study procedures did not involve changing the medication or the dose of the medication the participants were taking. Participants only changed the time they took their medications ( morning or evening). Questionnaires and check-in calls were used to assess for any adverse events.
Groups:
- Morning Group Medication Administration: Participants with Ulcerative Colitis taking Azathioprine or 6-Mercatopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Participants with Crohn's Disease taking Azathioprine or 6-Mercatopurine orally once a day. Dosage amount is per clinical care and not defined by the study protocol.
  Morning Group: Participants will take their IBD medication (either azathioprine or 6-mercaptopurine) between 6:00 am and 11:00 am.
Arm/Group | Evening Group Medication Administration | Morning Group Medication Administration
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/8
Other Adverse Events (participants affected / at risk) | 0/18 | 0/8

LIMITATIONS AND CAVEATS:
This was a single-center study with a limited number of IBD subjects that focused on metabolite levels and not clinical efficacy. Larger multicenter studies are needed since this was a "proof of concept" pilot study. Second, the overall dose of AZA/6-MP used in this study was low. Third, the study design relied on patient compliance with medication timing and circadian rhythms were assessed only by questionnaires.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT04304950/Prot_SAP_001.pdf
  • Informed Consent Form (2019-03-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT04304950/ICF_000.pdf